CLINICAL TRIAL: NCT03241719
Title: Novel Strategies to Improve Immunomodulation and Non-invasive Clinical Monitoring in Vascularized Composite Allotransplantation
Brief Title: Novel Strategies to Improve Immunomodulation and Non-invasive Clinical Monitoring in VCA
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants are currently receiving therapy under this protocol, funding is coming to an end and the PI is leaving the institution.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bodhan Pomahac, Director, Plastic Surgery Transplantation, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000590
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Amputation, Traumatic; Amputation;Traumatic;Old; Face Injury; Face; Deformity; Abdominal Wall Defect
MeSH Terms: conditions — Amputation, Traumatic; Facial Injuries; Facies; Congenital Abnormalities | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects who receive transplantation and undergo IL-2 treatment
  Interventions: Drug: IL-2

INTERVENTIONS:
Drug: IL-2 — Subjects will receive vascularized composite allotransplantation (e.g. facial, hand and/or abdominal wall transplants) under conventional immune suppression. No sooner than 3 months after VCA, subjects will receive a protocol of daily recombinant IL-2 at low doses for 8 weeks.

SUMMARY:
The objective of this study is to develop a feasible and safe regimen for minimization of immune suppression in recipients of vascularized composite allotransplants (VCA) using a daily dose of recombinant IL-2. In order to achieve this aim, this trial will:

1. Perform VCA in 5 eligible subjects;
2. Administer recombinant IL-2 at a low-dose to promote the expansion and function of regulatory T cells in subjects who received VCA; and
3. Minimize immune suppression to tacrolimus single therapy in subjects who received VCA and recombinant IL-2.

This trial will also investigate if it is possible to predict immune rejection in VCA using blood and tissue samples from recipients of VCA.

Lastly, this trial will develop non-invasive technologies to monitor for VCA rejection. These technologies will involve magnetic resonance imaging. Multi-contrast ultra-high resolution MR imaging (MRI) with serial direct planimetry will be performed in recipients of VCA.

ELIGIBILITY:
Inclusion Criteria:

For the VCA portion of the study:

* Patients referred due to one or more of these conditions: (1) severe facial deformity comprising more than 25% of the facial area and/or one or more of the central facial units (i.e. lip(s), nose, eye(s)), (2) single or bilateral upper limb(s) amputation, where at least one of the limbs was amputated at the level of the wrist or more proximal, up to the functional shoulder joint, and (3) severe abdominal wall defect comprising more than 50% of the functional abdominal wall.
* Injuries must have taken place no more than 15 years and no less than 6 months prior to presentation for consideration.
* All other conventional reconstruction approaches will have been either exhausted, or ruled out due to poor prognosis of outcomes.
* Patients will need to possess strong motivation and a willingness to commit to post-transplant rehabilitation.
* Normal renal and hepatic function within acceptable medical parameters

For the recombinant IL-2 phase of the study:

* At least 3 months have elapsed since the VCA transplant operation
* At least 4 weeks on stable immune suppression and steriods (<5 mg QD).
* No addition or subtraction of other immunosuppressive medications for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range for that drug.
* Medical evaluations, clinical and laboratory assessments must deem that participants have adequate organ function.
* The effects of some of the study drugs on the developing human fetus are unknown, or toxic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence prior to study entry and for the duration of study participation). Should a women become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Subjects must be able to understand and willing to sign a written informed consent document.
* Skin biopsies from the transplanted parts must show no evidence of rejection for at least 3 months prior to study enrollment.

Exclusion Criteria:

For the VCA portion of the study:

* History of poor compliance with prostheses or rehabilitation
* Impaired renal, cardiac and/or pulmonary function
* Compromised ability to understand the risk and benefits of participation in the study
* Active malignancy
* Single non-dominant upper limb amputation and no other vascularized composite tissue injuries justifying VCA

For the IL-2 portion of the study:

* Active infection
* Non-healing wounds
* Pregnancy, because of the potential for teratoenic or abortifacient effects. There is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother, therefore breastfeeding should be discontinued.
* Rejection episodes within the past 3 months
* Concurrent use of calcineurin-inhibitor plus sirolimus
* New immunosuppressive medication in the 4 weeks prior
* Post-transplant exposure to T-cell or IL-2 targeted medication (e.g. ATG, alemtuzumab, basiliximab, denileukin diftitox) within 100 days prior.
* Active malignant relapse
* Donor lymphocyte infusion within 100 days prior
* Inability to comply with IL-2 treatment regime
* HIV-positive individuals because of the potential for lethal infections.
* Other investigational drugs within 4 weeks prior to enrollment, unless cleared by the principal investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Number of regulatory T cells | 4-24 months

SECONDARY OUTCOMES:
Number of episodes of rejection | 1-24 months
T-cell alloreactivity measured by ELISPOT | 4-24 months
Steroid dose | 6-24 months
Mycophenolate dose | 8-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Pomahac, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No